CLINICAL TRIAL: NCT05429268
Title: A Phase 3, Single-Arm, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of Tafasitamab Plus Lenalidomide in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Study to Evaluate the Safety and Efficacy of Tafasitamab Plus Lenalidomide in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (firmMIND)
Acronym: firmMIND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMOR 0208-305; 2023-505579-53-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma
Keywords: MOR00208; INCMOR00208; tafasitamab; lenalidomide; firmMIND; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tafasitamab and Lenalidomide (Experimental): Tafasitamab and lenalidomide will be coadministered for up to 12 cycles (28 days per cycle).followed by tafasitamab monotherapy (in participants with stable disease or better) until treatment withdrawal criteria are met.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — Tafasitamab will be administered intravenously in 28-day cycles. During Cycles 1 through 3, tafasitamab will be administered weekly on Days 1, 8, 15, and 22; an additional loading dose will be administered on Cycle 1 Day 4. Starting with Cycle 4, tafasitamab will be administered on Days 1 and 15 of each cycle.
  Other Names: INCMOR00208; MOR00208
Drug: Lenalidomide — Participants will self-administer lenalidomide capsules orally on Days 1-21 of each 28-day cycle, up to 12 cycles.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of of tafasitamab plus lenalidomide in adults with diffuse large B-cell lymphoma (DLBCL) who have relapsed or are refractory to at least 1 but no more than 3 previous systemic DLBCL treatment regimens and who are not eligible for high-dose chemotherapy (HDC) and autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of any of the following:

  1. Diffuse large B-cell lymphoma not otherwise specified
  2. T cell/histiocyte-rich large B-cell lymphoma
  3. Epstein-Barr virus positive DLBCL of the elderly
  4. Grade 3b follicular lymphoma
  5. Composite lymphoma with a DLBCL component with a subsequent DLBCL relapse
  6. Evidence of histological transformation from an earlier diagnosis of low grade lymphoma (ie, an indolent pathology such as follicular lymphoma, marginal zone lymphoma, chronic lymphocytic leukemia) into DLBCL, with a subsequent DLBCL relapse
* Willingness to undergo tumor biopsy requirements for the study, (or have archival lymph node or tissue block from the most recent biopsy, not to exceed 3 years prior to C1D1).
* Willingness to undergo bone marrow biopsy/aspirate collections.
* History of relapsed/progressive/recurrent disease according to the International Working Group response criteria after the most recent systemic therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate hematologic, hepatic, and renal function,
* Left ventricular ejection fraction (LVEF) ≥ 50%,
* Willingness to avoid pregnancy or fathering children,

Exclusion Criteria:

* Any other histological type of lymphoma according to the WHO 2016 classification of lymphoid neoplasms, including:

  1. primary mediastinal (thymic) large B-cell lymphoma,
  2. Burkitt lymphoma,
  3. Primary refractory diffuse large B-cell lymphoma (DLBCL),
  4. History of double- or triple-hit DLBCL.
* Participants who, within 30 days prior to Cycle 1 Day 1, have:

  1. Not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma-specific therapy
  2. Undergone major surgery or suffered from significant traumatic injury
  3. Received live vaccines or have an anticipated need for such vaccination while receiving study treatment
  4. Required parenteral antimicrobial therapy for active, intercurrent infections
* Have undergone ASCT within the period ≤ 3 months prior to signing consent.
* Have undergone previous allogenic stem cell transplantation.
* Inadequate recovery (> Grade 1) from prior treatment toxicity and/or complications from major surgery before Cycle 1 Day 1.
* Have a history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or are at high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period.
* Prior history of malignancies other than DLBCL, unless disease-free for ≥ 5 years prior to screening.
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction, New York Heart Association Class II to IV congestive heart failure, uncontrolled arrhythmia, and/or cardiac conduction issues, within 6 months of Cycle 1 Day 1.
* Any of the following positive tests:

  1. Known seropositive for or history of active viral infection with HIV.
  2. Known positive test result for hepatitis C (HCV antibody serology testing) and a positive test result for HCV RNA.
  3. Known positive test results for chronic HBV infection (defined by HBsAg positivity). Participants with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA was undetectable

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 24 months
  Percentage of participants having best response of Complete Response (CR) or Partial Response (PR) as per Independent Review Committee and investigator's assessment.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Approximately 24 months
  Defined as the time from the first documented CR or PR until the date of first documented disease progression or death due to any cause, whichever occurs first, among participants who achieve CR or PR per Independent Review Committee (IRC) assessment and investigator's assessment.
Progression Free Survial (PFS) | Approximately 24 months
  Defined as the time from the date of first dose until the first documented disease progression, or death due to any cause, whichever occurs first per IRC assessment and investigator's assessment.
Disease Control Rate (DCR) | Approximately 24 months
  Defined as the percentage of participants who achieve CR, PR, or SD as per IRC assessment and investigator's assessment.
Time to Next Treatment (TTNT) | Approximately 24 months
  Defined as the time from first dose until the initiation of new anticancer therapy or death due to any reason, whichever occurs first.
Overall Survival (OS) | Approximately 24 months
  Defined as the time from the date of first dose until death due to any cause.
Number of treatment-emergent adverse events | Approximately 24 months
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study treatment up to 90 days after last dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Manzke, MD, Study Director — Incyte Corporation
Locations (61):
- Bulgaria (5):
  - Medical University Plovdiv, Plovdiv
  - Acibadem Cityclinica Mhat Tokuda, Sofia
  - Umhat Alexandrovska Sofia, Sofia
  - Umhat Sv. Ivan Rilski Ead, Sofia
  - Specialized Hospital For Active Treatment of Oncological Diseases - Sofia District Eood, Sofia
- Croatia (3):
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Merkur, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (2):
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice, Prague
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen, Debrecen
  - Markhot Ferenc Korhaz, Eger
  - Somogy Medyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Szeged
- Ireland (3):
  - Bon Secours Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Mc, Jerusalem
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kefar Sava
- Norway (2):
  - Akershus University Hospital, Lorenskog
  - Universitetssykehuset I Trondheim - St. Olavs Hospital, Trondheim
- Poland (8):
  - Szpital Uniwersytecki Nr 2 Im Dr. Jana Biziela, Bydgoszcz
  - Medical University of Gdansk, Gdansk
  - Szpital Morski Im. Pck Sp. Z O.O, Gdynia
  - University Public Hospital Nr 1, Lublin
  - Oddzia Kliniczny Hematologii, Olsztyn
  - Pratia Poznan, Skórzewo
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego, Wroclaw
- Romania (4):
  - Coltea Clinical Hospital, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
- Serbia (4):
  - Clinic For Hematology, University Clinical Center Serbia, Belgrade
  - Institute For Pulmonary Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinic of Hematology Clinical Center of Vojvodina, Novi Sad
- Turkey (Türkiye) (11):
  - Hacettepe University Cancer Institute Clinical Oncology Department, Ankara
  - Gazi University Hospital Gazi University Faculty of Medicine, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ozel Liv Hospital Onkoloji Klinigi, Ankara
  - Vkf American Hospital, Istanbul
  - Marmara Universitesi Pendik Egitim, Istanbul
  - Ege University Hospital, Izmir
  - Ercyes University Medical School, Kayseri
  - Tekrda-Nk Tp Fakltesi, Merkez
  - Mersin University Medical Faculty, Mersin
  - Dr. Abdurrahman Yurtaslan Onkology Teaching and Research Hospitalerciyes Universitesi Tip Faklutesi, Yenimahalle
- United Kingdom (2):
  - Antrim Area Hospital Northern Health Social Care Trust, Antrim
  - Belfast Health and Social Care Trust, of Trust Headquarters, Belfast

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to Evaluate the Safety and Efficacy of Tafasitamab Plus Lenalidomide in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (firmMIND) — https://incyteclinicaltrials.com/studies/incmor-0208-305